CLINICAL TRIAL: NCT07215065
Title: Examining Heavy Metal Exposure and Respiratory Health in Young Adult Electronic Cigarette Users
Status: Recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Alayna Tackett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-25119; NCI-2025-06572 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-10-08; First posted 2025-10-10 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Heavy Metal Exposure From Vaping

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Participants vape their own electronic cigarette device as much or as little as they like over 30 minutes on study. Participants also undergo saliva sample collection, spirometry to measure respiratory function, and complete questionnaires.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study
  Other Names: Non-Interventional Observational Study

SUMMARY:
This study investigates heavy metal exposure in young adults who use electronic cigarettes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify and quantify heavy metals (HM) concentration in the saliva of e-cigarette users.

II. Examine changes in pulmonary functioning and HM concentration pre/post vaping.

III. Examine the association between vaping intensity and HM concentration in the saliva of e-cigarette users.

OUTLINE: This is an observational study.

Participants vape their own electronic cigarette device as much or as little as they like over 30 minutes on study. Participants also undergo saliva sample collection, spirometry to measure respiratory function, and complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-29 years
* Established electronic cigarette (EC) user (participant uses ECs on a daily/weekly basis [used on ≥ 5 days in past 30-days] for the past 3 months)
* Willing to abstain from nicotine for at least 12 hours before the laboratory visit
* Willing to not eat food or drink water/beverages for at least 30 minutes before the laboratory visit [required for salivary collection]
* Utilize 4th generation EC products (pod-mod or disposable EC products; e.g., JUUL, Hyde)
* Must be able to read and write in English

Exclusion Criteria:

* Recently COVID-19+ (defined as a positive test in the past 30 days) or a recent COVID-19 hospitalization (within the past 6 months)
* Attempting to quit the use of ECs
* Past 30-day use of other tobacco products (e.g., combustible cigarettes)
* Is pregnant, planning on becoming pregnant and/or breastfeeding [will be verified using a urine pregnancy test]
* Self-reported severe or significant psychological and/or psychiatric conditions [e.g., not currently receiving treatment/medication; only past and/or stable conditions will be allowed]
* A history of cardiac events and/or distress within the past 3 months
* Diagnosed with a chronic, serious lung disease or current infection (e.g., pneumonia, pulmonary edema)
* Are deaf, hard of hearing, or have a severe motor disability

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults (aged 18 - 29 years) who are established and current EC users.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Heavy metal concentration in the saliva of e-cigarette users | Baseline, Immediately Following Vaping Session
  Identify and quantify HM concentrations in the saliva among all participants in the sample before and after their 30 minute vaping session.
Spirometry to Measure the Change From Baseline in Forced Vital Capacity (FVC) | Baseline, Immediately Following Vaping Session
  Participants will complete spirometry (a pulmonary function test) before and immediately after the completion of the 30 minute vaping session.
Spirometry to Measure the Change From Baseline in Forced Expiratory Volume in One Second (FEV1) | Baseline, Immediately Following Vaping Session
  Participants will complete spirometry (a pulmonary function test) before and immediately after the completion of the 30 minute vaping session.
E-cigarette puffing behavior | Up to 30 minutes
  E-cigarette puffing behavior will be measured with a topography device that records frequency, duration, and flow rate of e-cigarette puffs. These measures are combined to inform the overall measure of e-cigarette puffing behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Alayna P Tackett, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu